CLINICAL TRIAL: NCT06114992
Title: Servo-n High-Frequency Oscillatory Ventilation in Clinical Practice: A Prospective, Observational, Single-arm and Multi-center Study
Brief Title: Servo-n HFOV Study: Safety and Performance in Neonates and Infants
Status: Recruiting | Type: Observational
Sponsor: Maquet Critical Care AB (Industry)
Collaborators: NAMSA (Other); Paediatric and Neonatal Mechanical Ventilation (PNV) Consulting (Unknown)
Responsible Party: Sponsor
Other Study IDs: EVU-215176
Record Dates: First submitted 2023-10-11; First posted 2023-11-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Elective HFOV for Respiratory Failure in Neonates/Infants; Rescue HFOV in Neonates and/Infants With Refractory Respiratory Failure Under Conventional Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 120 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Servo-n HFOV treatment: As this study is single-armed (non-controlled), all patients in this study receive the same treatment, i.e. Servo-n HFOV treatment. There are however two subgroups, elective HFOV and rescue HFOV treatment
  Interventions: Device: Servo-n HFOV modes

INTERVENTIONS:
Device: Servo-n HFOV modes — Treatment with high frequency oscillatory ventilation with Servo-n device in accordance to Standard of Care

SUMMARY:
The purpose of this study is to evaluate the safety and performance of High-Frequency Oscillatory Ventilation (HFOV) modes of the Servo-n ventilator in neonates and infants, by using a prospective, observational, single-arm (i.e., non-controlled) and multi-center Post-Market Follow-up (PMCF) study design. HFOV treatment will be evaluated by assessing ventilation and oxygenation variables, and safety will be evaluated by documentation of device related adverse events.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and performance of HFOV modes of the Servo-n ventilator in neonates and infants. This is a prospective, observational, single-arm (i.e., non-controlled) and multi-center PMCF study in neonates and infants between 0.3 to 8 kg. All study procedures are within each hospital's routine clinical practice.The primary endpoints includes variables which are routinely used per clinical practice for assessing the status of patient's ventilation and oxygenation, respectively. Secondary endpoints are used to evaluate safety of Servo-n HFOV during its use by assessing rates of adverse event/ device deficiencies related to the Servo-n HFOV device, and by assessing rates of mortality, Bronchopulmonary Dysplasia (BPD) and Retinopathy at Intensive Care Unit (ICU) discharge. Data collection will take place up to 24 hours prior to HFOV treatment, during HFOV and up to ICU discharge. Additional general data such as ventilator settings, reasons for initiating/terminating HFOV treatment and demographics will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent by the patient's legally designated representative(s) (may be obtained as deferred consent up to 24 hours after HFOV initiation: valid for both elective and rescue HFOV patients)
* Patients eligible for HFOV ventilation with Servo-n:

  * Patient is either switched from conventional mechanical ventilation or HFOV with other device to Servo-n HFOV based on clinicians judgement (rescue HFOV). Note: the reason for the switch has to be that the patient failed to oxygenate or ventilate adequately with CMV or the other HFOV device

    ; OR
  * Patient was prior without or with any type of non-invasive respiratory support and is put on invasive HFOV treatment based on clinicians judgement (elective HFOV)
* Patient has not already been on HFOV in a previous episode, unless the etiology of respiratory failure has changed during the same hospitalisation. For example, initial HFOV treatment for RDS, second HFOV episode of NARDS of any etiology (will be enrolled as a new patient case). NOTE1: When a patient failed weaning on conventional ventilation within 6 hours, requiring to be put back on HFOV it will be counted as one HFOV episode (weaning failure) NOTE2: When a patient is temporarily put on conventional ventilation for transport or a surgical intervention, and will be put back to HFOV afterwards, it will be counted as one HFOV episode (HFOV paused).
* Patient has a body weight from 0.3 to 8.0 kg

Exclusion Criteria:

* Diagnosis of congenital diaphragmatic hernia
* Severe cardiac anomaly expected to need corrective surgery or catheter-based intervention within 30 days from birth
* Cyanotic heart disease
* Intracranial hemorrhage, Grade III or IV
* Congenital malformations with the exception of isolated lung hypoplasia
* Persistent pulmonary hypertension (PPHN) with a documented shunt on the level of the foramen ovale
* Bronchopulmonary Dysplasia (BPD) /Chronic Lung Disease (CLD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both preterm and term (0.3-8 kg) neonatal/infant patient group requiring HFOV treatment. Subjects on elective HFOV and rescue HFOV, will be enrolled from up to 10 sites in European countries.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects that achieved and/or maintained target ranges for oxygenation, as measured by preductal Saturation of Peripheral Oxygen (SpO2). | After Servo-n HFOV treatment, expected treatment duration 1-30 days
  Oxygenation response, elective HFOV patients
Proportion of subjects that achieved and/or maintained target ranges for ventilation as measured either by Partial Pressure of Carbon Dioxide (PCO2) (if available blood gas) or Transcutaneous Carbon Dioxide (TcCO2) | After Servo-n HFOV treatment, expected treatment duration 1-30 days
  Ventilation response, elective HFOV patients
Proportion of subjects that maintained or improved values for oxygenation as measured by the SpO2/FiO2 ratio and/ or achieved target ranges for oxygenation (preductal SpO2) | After Servo-n HFOV treatment, expected treatment duration 1-30 days
  Oxygenation response, rescue HFOV patients
Proportion of subjects that maintained or improved values, and/or achieved target ranges, for ventilation as measured either by PCO2 (if available blood gas) or TcCO2. | After Servo-n HFOV treatment, expected treatment duration 1-30 days
  Ventilation response, rescue HFOV patients

SECONDARY OUTCOMES:
The occurrence of reported Servo-n HFOV device (including accessories) deficiencies and adverse device effects and serious adverse device effects (ADE and SADE) | After Servo-n HFOV treatment, expected treatment duration 1-30 days
  Device deficiencies and adverse events
Patient outcome at ICU discharge | Through study completion (at ICU discharge), expected up to 120 days
  Events to be noted are: death caused by respiratory failure, death caused by circulatory failure, all-cause death, device related death, retinopathy and bronchopulmonary dysplasia
Assessment of oxygenation status | From available blood gas and at Baseline (-4h -2h, -1h, 0h), During HFOV (0h, 30min, 1h, 2h, 4h, 6h. etc every 6 h), Post HFOV (2h, 4h, 6h, 12h and 24h)
  Oxygen Saturation (SO2)
Assessment of ventilation status | From available blood gas and at Baseline (-4h -2h, -1h, 0h), During HFOV (0h, 30min, 1h, 2h, 4h, 6h. etc every 6 h), Post HFOV (2h, 4h, 6h, 12h and 24h)
  Partial pressure of CO2 (PCO2)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rimensberger, Prof. MD, Study Chair — PNV consulting
Locations (4):
- France (2):
  - CHU Montpellier-Arnaud de Villeneuve, Montpellier
  - Antoine-Béclère Hospital, Paris
- Poznan University of Medical Sciences, Poznan, Poland
- University Hospital of Geneva (HUG),, Geneva, Switzerland